CLINICAL TRIAL: NCT01137006
Title: An Open-Label, Dose-Escalation Phase 1/1b Study of the Anti-gp75 Monoclonal Antibody IMC-20D7S In Patients With Malignant Melanoma Who Have Progressed After or During at Least One Treatment With Standard Cytotoxic Treatment or/and Immunotherapy Therapy or For Whom Standard Therapy is Not Indicated
Brief Title: An Open-Label, Dose-Escalation Study of IMC-20D7S In Participants With Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13945; CP22-0901 (Other: ImClone, LLC); I4Z-IE-JDEA (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Malignant Melanoma
Keywords: Melanoma; Phase I; antibody; melanin; tyrosinase related protein 1; glycoprotein; 20D7S
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMC-20D7S (1A-4A Cohorts) (Experimental): Escalating doses up to 30 milligrams per kilogram (mg/kg) administered intravenously (i.v.) every 2 weeks; includes Cohorts 1A, 2A, 3A, and 4A.
  Interventions: Biological: IMC-20D7S (Cohort 1A); Biological: IMC-20D7S (Cohort 2A); Biological: IMC-20D7S (Cohort 3A); Biological: IMC-20D7S (Cohort 4A)
- IMC-20D7S (1B-3B Cohorts) (Experimental): Escalating doses up to 30 mg/kg administered i.v. every 3 weeks; includes Cohorts 1B, 2B, and 3B.
  Interventions: Biological: IMC-20D7S (Cohort 1B); Biological: IMC-20D7S (Cohort 2B); Biological: IMC-20D7S (Cohort 3B)

INTERVENTIONS:
Biological: IMC-20D7S (Cohort 1A) — 5 mg/kg i.v. every 2 weeks.
  Administered every other week on Days 1 and 15 of each treatment cycle.
  If no dose-limiting toxicity (DLT) in first 3 participants or 1 DLT in 6 participants, then enrollment into Cohort 2A.
  Other Names: LY3012215
  Arms: IMC-20D7S (1A-4A Cohorts)
Biological: IMC-20D7S (Cohort 2A) — 10 mg/kg i.v. every 2 weeks.
  Administered every other week on Days 1 and 15 of each treatment cycle.
  If no DLT in first 3 participants or 1 DLT in 6 participants in Cohort 2A, then enrollment into Cohort 3A.
  Other Names: LY3012215
  Arms: IMC-20D7S (1A-4A Cohorts)
Biological: IMC-20D7S (Cohort 3A) — 20 mg/kg i.v. every 2 weeks.
  Administered every other week on Days 1 and 15 of each treatment cycle.
  If no DLT in first 3 participants or 1 DLT in 6 participants in Cohort 3A, then enrollment into Cohort 4A.
  Other Names: LY3012215
  Arms: IMC-20D7S (1A-4A Cohorts)
Biological: IMC-20D7S (Cohort 4A) — 30 mg/kg i.v. every 2 weeks.
  Administered every other week on Days 1 and 15 of each treatment cycle.
  Other Names: LY3012215
  Arms: IMC-20D7S (1A-4A Cohorts)
Biological: IMC-20D7S (Cohort 1B) — 10 mg/kg i.v. every 3 weeks.
  Administered every 3 weeks on Days 1 and 22 of each treatment cycle.
  If no dose-limiting toxicity (DLT) in first 3 participants or 1 DLT in 6 participants in Cohort 1B, then enrollment into Cohort 2B.
  Other Names: LY3012215
  Arms: IMC-20D7S (1B-3B Cohorts)
Biological: IMC-20D7S (Cohort 2B) — 20 mg/kg i.v. every 3 weeks.
  Administered every 3 weeks on Days 1 and 22 of each treatment cycle.
  If no DLT in first 3 participants or 1 DLT in 6 participants in Cohort 2B, then enrollment into Cohort 3B.
  Other Names: LY3012215
  Arms: IMC-20D7S (1B-3B Cohorts)
Biological: IMC-20D7S (Cohort 3B) — 30 mg/kg i.v. every 3 weeks.
  Administered every 3 weeks on Days 1 and 22 of each treatment cycle.
  Other Names: LY3012215
  Arms: IMC-20D7S (1B-3B Cohorts)

SUMMARY:
A dose-escalation study designed to determine the safety, maximum tolerated dose (MTD), anti-melanoma activity, antibody blood levels and progression-free survival (PFS) in participants with malignant melanoma receiving IMC-20D7S either every 2 weeks or every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically or cytologically confirmed cutaneous, mucosal, or uveal malignant melanoma which has progressed after or during at least 1 treatment with standard cytotoxic treatment or/and immunotherapy [for example (e.g.), treatment with cytokines, monoclonal antibodies, and vaccines] and is not regarded to be a candidate for a potentially curative, higher priority treatment for melanoma
* Participant is ≥18 years of age
* Participant has either measurable disease as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) or evaluable disease
* At least 21 days must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent or device, or prior radiation therapy. Relative to participant's treatment with non-approved biological products (eg, monoclonal antibodies), a minimum of 2 half-lives must have passed for eligibility to be considered
* Participant has resolution of all clinically significant toxic effects of prior cancer therapy to Grade ≤1 according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.02 (NCI-CTCAE v4.02)
* Participant has adequate hematological function, hepatic function, and renal function

Exclusion Criteria:

* Participant has undergone major surgery [e.g., laparotomy, thoracotomy, removal of organ(s)] within 21 days prior to study entry
* Participant has elective or planned surgery to be conducted during the trial
* Participant has documented and/or symptomatic brain or leptomeningeal metastases
* Participant is receiving systemic steroids or other immunosuppressive medications. (Intermittent use of steroid-containing medications e.g., for asthma exacerbation or for skin lesions is permitted)
* Participant has an uncontrolled undercurrent illness
* Participant has a concurrent active malignancy other than adequately treated nonmelanomatous skin cancer or other noninvasive carcinoma or in situ neoplasm
* Participant has a known allergy to any of the treatment components (monoclonal antibodies or other therapeutic proteins such as fresh frozen plasma, human serum albumin, cytokines, or interleukins). In the event that there is suspicion the participant may have allergies, the participant should be excluded
* Participant is pregnant or lactating
* Participant has known human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - ImClone Investigational Site, Boston, Massachusetts
  - ImClone Investigational Site, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A completed participant (pt) finished the first 4 or 6 weeks of therapy or discontinued due to toxicity. Cohort (C)1A pts were treated sequentially. The next cohort started when all pts finished Cycle 1 of current cohort. Cohorts 1B-3B started if supported by C1A and C2A pharmacokinetic (PK) data and if maximum tolerated dose (MTD) not established.
Groups:
- Cohort 1A (5 mg/kg, q2w): IMC-20D7S: 5 milligrams per kilogram (mg/kg) IMC-20D7S administered intravenously (i.v.) as an infusion every other week (q2w) on Days 1 and 15 of each 4-week treatment cycle until disease progression, unacceptable toxicity, or other withdrawal criteria were met. There were ≥7 days between the start of treatment for each participant in this cohort.
- Cohort 2A (10 mg/kg, q2w): IMC-20D7S: 10 mg/kg IMC-20D7S administered i.v. as an infusion q2w on Days 1 and 15 of each 4-week treatment cycle until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- Cohort 3A (20 mg/kg, q2w): IMC-20D7S: 20 mg/kg IMC-20D7S administered i.v. as an infusion q2w on Days 1 and 15 of each 4-week treatment cycle until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- Cohort 4A (30 mg/kg, q2w): IMC-20D7S: 30 mg/kg IMC-20D7S administered i.v. as an infusion q2w on Days 1 and 15 of each 4-week treatment cycle until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- Cohort 1B (10 mg/kg, q3w): IMC-20D7S: 10 mg/kg IMC-20D7S administered i.v. as an infusion every three weeks (q3w) on Days 1 and 22 of each 6-week treatment cycle until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- Cohort 2B (20 mg/kg, q3w): IMC-20D7S: 20 mg/kg IMC-20D7S administered i.v. as an infusion q3w on Days 1 and 22 of each 6-week treatment cycle until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- Cohort 3B (30 mg/kg, q3w): IMC-20D7S: 30 mg/kg IMC-20D7S administered i.v. as an infusion q3w on Days 1 and 22 of each 6-week treatment cycle until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
Period: Overall Study
Arm/Group | Cohort 1A (5 mg/kg, q2w) | Cohort 2A (10 mg/kg, q2w) | Cohort 3A (20 mg/kg, q2w) | Cohort 4A (30 mg/kg, q2w) | Cohort 1B (10 mg/kg, q3w) | Cohort 2B (20 mg/kg, q3w) | Cohort 3B (30 mg/kg, q3w)
Started | 3 | 3 | 8 | 3 | 3 | 4 | 3
Completed at Least 1 Treatment Cycle | 3 | 3 | 8 | 3 | 3 | 4 | 3
Completed | 3 | 3 | 8 | 3 | 3 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received any amount of IMC-20D7S.
Groups:
- Cohort 1A (5 mg/kg, q2w): IMC-20D7S: 5 mg/kg IMC-20D7S administered i.v. as an infusion q2w on Days 1 and 15 of each 4-week treatment cycle until disease progression, unacceptable toxicity, or other withdrawal criteria were met. There were ≥7 days between the start of treatment for each participant in this cohort.
- Cohort 1B (10 mg/kg, q3w): IMC-20D7S: 10 mg/kg IMC-20D7S administered i.v. as an infusion q3w on Days 1 and 22 of each 6-week treatment cycle until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- Total: Total of all reporting groups
Arm/Group | Cohort 1A (5 mg/kg, q2w) | Cohort 2A (10 mg/kg, q2w) | Cohort 3A (20 mg/kg, q2w) | Cohort 4A (30 mg/kg, q2w) | Cohort 1B (10 mg/kg, q3w) | Cohort 2B (20 mg/kg, q3w) | Cohort 3B (30 mg/kg, q3w) | Total
Number analyzed (Participants) | 3 | 3 | 8 | 3 | 3 | 4 | 3 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.7 (5.50) | 64.9 (4.92) | 69.8 (8.37) | 61.1 (11.70) | 66.6 (4.41) | 69.1 (5.53) | 65.4 (18.90) | 68.2 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 1 | 1 | 1 | 2 | 11
  Male | 1 | 2 | 5 | 2 | 2 | 3 | 1 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 7 | 3 | 3 | 4 | 3 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 2 | 2 | 8 | 3 | 3 | 4 | 3 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 8 | 3 | 3 | 4 | 3 | 27

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of IMC-20D7S
Description: The MTD was defined as the dose preceding the dose level at which 2 participants experienced a dose-limiting toxicity (DLT) during treatment Cycle 1. A DLT was defined as any Grade 3 or above toxicity that emerged during study treatment and was clearly not attributable to malignant melanoma or co-medication and was possibly, probably, or definitely related to IMC-20D7S in the judgment of the investigator. No DLT was observed in the study; a provisional MTD was established.
Time Frame: Baseline to toxicity [up to end of Cycle 1 (4 or 6-week cycles)]
Population: Participants who completed Cycle 1 of treatment.
Measure: Number; unit: mg/kg q2w
Groups:
- IMC-20D7S: IMC-20D7S: Escalating doses (up to 30 mg/kg IMC-20D7S) administered i.v. as an infusion either q2w on Days 1 and 15 of each 4-week treatment cycle or q3w on Days 1 and 22 of each 6-week treatment cycle.
  Treatment continued until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
Arm/Group | IMC-20D7S
Number analyzed (Participants) | 27
mg/kg q2w | 20

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), Other Non-Serious Adverse Events (AEs), or Death
Description: A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Baseline through 30 days post last dose (up to 31 weeks)
Population: Participants who received any amount of IMC-20D7S .
Measure: Number; unit: participants
Arm/Group | Cohort 1A (5 mg/kg, q2w) | Cohort 2A (10 mg/kg, q2w) | Cohort 3A (20 mg/kg, q2w) | Cohort 4A (30 mg/kg, q2w) | Cohort 1B (10 mg/kg, q3w) | Cohort 2B (20 mg/kg, q3w) | Cohort 3B (30 mg/kg, q3w)
Number analyzed (Participants) | 3 | 3 | 8 | 3 | 3 | 4 | 3
participants
  SAEs | 1 | 1 | 5 | 2 | 0 | 4 | 0
  Other Non-Serious AEs | 3 | 3 | 8 | 3 | 2 | 4 | 3
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: IMC-20D7S Pharmacokinetics (PK): Maximum Concentration (Cmax)
Description: A non-validated assay was used to determine individual serum concentrations of IMC-20D7S. Thus, analyses of PK data were not conducted.
Time Frame: Cycles 1 and 3: Prior to, immediately after, and 0.5, 1, 2, 4, 8, 24, 48 (Cycle 3 only), 96, 168, 240, and 336 hours (h) post first infusion. Cycles 2 and 4: Prior to and 1 h post first infusion.
Population: No participant was analyzed.
Arm/Group | Cohort 1A (5 mg/kg, q2w) | Cohort 2A (10 mg/kg, q2w) | Cohort 3A (20 mg/kg, q2w) | Cohort 4A (30 mg/kg, q2w) | Cohort 1B (10 mg/kg, q3w) | Cohort 2B (20 mg/kg, q3w) | Cohort 3B (30 mg/kg, q3w)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: IMC-20D7S PK: Minimal Concentration (Cmin)
Description: as for outcome 3
Time Frame: Cycles 1 and 3: Prior to, immediately after, and 0.5, 1, 2, 4, 8, 24, 48 (Cycle 3 only), 96, 168, 240, and 336 h post first infusion. Cycles 2 and 4: Prior to and 1 h post first infusion.
Population: No participant was analyzed.
Arm/Group | Cohort 1A (5 mg/kg, q2w) | Cohort 2A (10 mg/kg, q2w) | Cohort 3A (20 mg/kg, q2w) | Cohort 4A (30 mg/kg, q2w) | Cohort 1B (10 mg/kg, q3w) | Cohort 2B (20 mg/kg, q3w) | Cohort 3B (30 mg/kg, q3w)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: IMC-20D7S PK: Half-life (t½)
Description: as for outcome 3
Time Frame: as for outcome 4
Population: No participant was analyzed.
Arm/Group | Cohort 1A (5 mg/kg, q2w) | Cohort 2A (10 mg/kg, q2w) | Cohort 3A (20 mg/kg, q2w) | Cohort 4A (30 mg/kg, q2w) | Cohort 1B (10 mg/kg, q3w) | Cohort 2B (20 mg/kg, q3w) | Cohort 3B (30 mg/kg, q3w)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: IMC-20D7S PK: Clearance (Cl)
Description: as for outcome 3
Time Frame: as for outcome 4
Population: No participant was analyzed.
Arm/Group | Cohort 1A (5 mg/kg, q2w) | Cohort 2A (10 mg/kg, q2w) | Cohort 3A (20 mg/kg, q2w) | Cohort 4A (30 mg/kg, q2w) | Cohort 1B (10 mg/kg, q3w) | Cohort 2B (20 mg/kg, q3w) | Cohort 3B (30 mg/kg, q3w)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: IMC-20D7S PK: Area Under the Concentration Versus Time Curve (AUC)
Description: as for outcome 3
Time Frame: as for outcome 4
Population: No participant was analyzed.
Arm/Group | Cohort 1A (5 mg/kg, q2w) | Cohort 2A (10 mg/kg, q2w) | Cohort 3A (20 mg/kg, q2w) | Cohort 4A (30 mg/kg, q2w) | Cohort 1B (10 mg/kg, q3w) | Cohort 2B (20 mg/kg, q3w) | Cohort 3B (30 mg/kg, q3w)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: IMC-20D7S PK: Volume of Distribution (Vd) at Steady State
Description: as for outcome 3
Time Frame: as for outcome 4
Population: No participant was analyzed.
Arm/Group | Cohort 1A (5 mg/kg, q2w) | Cohort 2A (10 mg/kg, q2w) | Cohort 3A (20 mg/kg, q2w) | Cohort 4A (30 mg/kg, q2w) | Cohort 1B (10 mg/kg, q3w) | Cohort 2B (20 mg/kg, q3w) | Cohort 3B (30 mg/kg, q3w)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants Who Develop Antibodies Against IMC-20D7S (Immunogenicity)
Description: Planned analyses for immunogenicity were not completed. A decision was made not to develop a validated immunogenicity assay because of the exploratory nature of the study and the analyses.
Time Frame: Prior to the first and second infusion in each cycle up to Cycle 7 (4- and 6-week cycles)
Population: No participant was analyzed.
Arm/Group | Cohort 1A (5 mg/kg, q2w) | Cohort 2A (10 mg/kg, q2w) | Cohort 3A (20 mg/kg, q2w) | Cohort 4A (30 mg/kg, q2w) | Cohort 1B (10 mg/kg, q3w) | Cohort 2B (20 mg/kg, q3w) | Cohort 3B (30 mg/kg, q3w)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was determined for participants who went beyond their first disease assessment and completed at least 1 treatment beyond Week 1 of treatment Cycle 3.
Time Frame: First dose to disease progression or death (up to 27 weeks)
Population: Participants who went beyond their first disease assessment and completed at least one treatment beyond Week 1 of treatment Cycle 3.
Measure: Number; unit: participants
Arm/Group | Cohort 1A (5 mg/kg, q2w) | Cohort 2A (10 mg/kg, q2w) | Cohort 3A (20 mg/kg, q2w) | Cohort 4A (30 mg/kg, q2w) | Cohort 1B (10 mg/kg, q3w) | Cohort 2B (20 mg/kg, q3w) | Cohort 3B (30 mg/kg, q3w)
Number analyzed (Participants) | 3 | 3 | 8 | 3 | 3 | 4 | 3
participants | 0 | 3 | 2 | 1 | 1 | 1 | 2

11. Secondary Outcome: Recommend Doses for Phase 2/3 Studies Based on MTD
Description: It was decided for administrative reasons to discontinue dosing at the provisional MTD rather than progress to Phase 1b.
Time Frame: Baseline to toxicity [up to end of Cycle 1 (4-or 6-week cycles)]
Population: No participant was analyzed.
Arm/Group | IMC-20D7S
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Cohort 1A (5 mg/kg, q2w) | Cohort 2A (10 mg/kg, q2w) | Cohort 3A (20 mg/kg, q2w) | Cohort 4A (30 mg/kg, q2w) | Cohort 1B (10 mg/kg, q3w) | Cohort 2B (20 mg/kg, q3w) | Cohort 3B (30 mg/kg, q3w)
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 5/8 | 2/3 | 0/3 | 4/4 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 8/8 | 3/3 | 2/3 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1A (5 mg/kg, q2w) (N=3) | Cohort 2A (10 mg/kg, q2w) (N=3) | Cohort 3A (20 mg/kg, q2w) (N=8) | Cohort 4A (30 mg/kg, q2w) (N=3) | Cohort 1B (10 mg/kg, q3w) (N=3) | Cohort 2B (20 mg/kg, q3w) (N=4) | Cohort 3B (30 mg/kg, q3w) (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1A (5 mg/kg, q2w) (N=3) | Cohort 2A (10 mg/kg, q2w) (N=3) | Cohort 3A (20 mg/kg, q2w) (N=8) | Cohort 4A (30 mg/kg, q2w) (N=3) | Cohort 1B (10 mg/kg, q3w) (N=3) | Cohort 2B (20 mg/kg, q3w) (N=4) | Cohort 3B (30 mg/kg, q3w) (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breath odour (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 4 (5) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (4) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile oedema (Reproductive system and breast disorders) | 0/1 (0) | 0/2 (0) | 0/5 (0) | 1/2 (1) | 0/2 (0) | 0/3 (0) | 0/1 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0/1 (0) | 0/2 (0) | 0/5 (0) | 1/2 (1) | 0/2 (0) | 0/3 (0) | 0/1 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.